CLINICAL TRIAL: NCT04805151
Title: Polypharmacy, Medication Appropriateness, Risk Factors, Clinical Outcomes and Predication on Medication Related Harm Post- Discharge From a Hospital for Surgical Patients
Brief Title: Polypharmacy and Associated Risk Factors and Clinical Outcomes for Surgical Patients Discharged From Hospital
Status: Active, not recruiting | Type: Observational
Sponsor: University of Iceland (Other)
Collaborators: Landspitali University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UI- 2021 polypharmacy
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Polypharmacy; General Surgery
Keywords: Polypharmacy; Potentially inappropriate medication list; Drug-related side effects and adverse reaction; Readmission; Patient discharge; Prediction tool; Start and stop; Inappropriate Prescribing; General surgery; Beers criteria; STOPP START criteria
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The World Health Organisation Patient Safety Challenge: Medication Without Harm has brought our attention to the importance of medication-related harm as a global public health issue. One of the major contributing factors is polypharmacy, the usage of multiple medicines at the same time. People are getting older and living longer with chronic diseases; they need more medications, which frequently leads to polypharmacy. Subsequently, they are at more risk of medication-related harm. The planned project is an epidemiological study on polypharmacy, medication appropriateness, risk factors, and clinical outcomes post-discharge from a hospital for surgical patients.

The study group hypothesise that pre-and post-operative polypharmacy and potentially inappropriate prescribing is common, especially among older patients, patients with a high comorbidity and frailty burden, and patients undergoing more complicated surgery. Our hypothesis is additionally that preoperative polypharmacy and potentially inappropriate prescribing is associated with a higher short- and long-term mortality, a longer primary hospitalization length of stay, and a higher risk of readmission.

DETAILED DESCRIPTION:
This is an observational, retrospective, single centered study, using clinical data from the patient's medical record from the hospital, the national prescription database of the Directorate of Health, and the and ICD-10 codes from primary care records. For this analysis, medicines will be classified into drug classes based on the first five characters of their WHO Anatomical Therapeutic Chemical (ATC) code. The prevalence (pre) and incidence (post) of polypharmacy (≥5 or more regular medicines) and hyper-polypharmacy (≥10 regular medicines) will be calculated. Potentially inappropriate prescribing will be assessed in individuals ≥65 years applying Beers 2019, Start and Stopp 2014, explicit prescribing criteria. The analysis will be restricted to older individuals, as Beers criteria have not been validated in younger age groups. The anticholinergic burden will be assessed for all individuals ≥18 years will be assessed by applying the anticholinergic burden scale This stratification is important in order to deliver targeted interventions in resource-limited healthcare settings

ELIGIBILITY:
Inclusion Criteria:

* Participants: surgery patients ≥18 years in admitted to Landspitali University Hospital over the period 2010-2018.

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is surgical patients in hospital settings. The cohort will include 100% of tertiary care surgical admissions in Iceland and 70-80% of secondary care in Iceland. The study population includes 56.000 number of participants.
Sampling Method: Probability Sample
Enrollment: 56000 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2024-06-02 (Estimated); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
Polypharmacy | 2010-2018
  Prevalence of polypharmacy (≥5 or more regular medicines) and hyper-polypharmacy (≥10 regular medicines) pre-admission and prevalence and incidence post-discharge for surgery patients ≥18 years in Iceland

SECONDARY OUTCOMES:
Clinical variables associated with the prevalence and incidence of polypharmacy | 2010-2018
  Clinical variables associated with the prevalence and incidence of polypharmacy and hyper-polypharmacy for the surgery patients ≥18 years in Iceland.
  Prevalence of potentially inappropriate prescribing amongst patients ≥65 years in Iceland by applying Beers 2019 and Start and Stopp explicit prescribing criteria. To investigate the association of potentially inappropriate prescribing with polypharmacy, patient-specific factors, drug classes, and outcomes.
  Prevalence of anticholinergic burden by applying the Anticholinergic burden scale in individuals aged ≥18 years in Iceland and investigate the association of anticholinergic burden with polypharmacy, patient-specific factors, drug classes (ACD-codes), and selected outcomes (temporary admission, long-term mortality, time to readmission)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sigurdsson, MD PhD, Principal Investigator — University of Iceland
Locations (1):
- Faculty of Pharmaceutical Sciences, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jonsdottir F, Blondal AB, Guethmundsson A, Bates I, Stevenson JM, Sigurethsson MI. Epidemiology and association with outcomes of polypharmacy in patients undergoing surgery: retrospective, population-based cohort study. BJS Open. 2023 May 5;7(3):zrad041. doi: 10.1093/bjsopen/zrad041. PMID 37194458